CLINICAL TRIAL: NCT03383003
Title: Comparison of Two Novel First-line Anti-Helicobacter Pylori Therapy: A Prospective Randomized Trial
Brief Title: Comparison of Two Novel First-line Anti-Helicobacter Pylori Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Tai M.D., Associate professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRMG8E1281
Record Dates: First submitted 2017-12-17; First posted 2017-12-26 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2017-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori eradication; High dose proton pump inhibitor; High dose Amoxicillin; Concomitant therapy
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose dual therapy (Experimental): Esomeprezole (Nexium)40 mg tid. and amoxicillin (Amolin) 750 mg qid. for 14 days
  Interventions: Drug: Nexium; Drug: Amolin
- Non-bismuth quadruple therapy (Active Comparator): Esomeprezole (Nexium) 40 mg bid.,clarithromycin (Klaricid) 500 mg bid., amoxicillin (Amolin) 1 g bid. and metronidazole (Flagyl) 500 mg bid. for 7 days
  Interventions: Drug: Nexium; Drug: Amolin; Drug: Klaricid; Drug: Flagyl

INTERVENTIONS:
Drug: Nexium — Esomeprazole ( Nexium )40 mg tid daily for 14 days in the high dose dual therapyarm and 40 mg bid daily for 7 days in the non-bismuth quadruple therapy
  Other Names: Esomeprazole
Drug: Amolin — Amoxicillin 750 mg qid daily for 14 days in the high dose dual therapy and amoxicillin 1 g bid daily for 7 days in the non-bismuth quadruple therapy
  Other Names: Amoxicillin
Drug: Klaricid — clarithromycin 500 mg bid daily for 7 days in the non-bismuth quadruple therapy
  Other Names: Clarithromycin
  Arms: Non-bismuth quadruple therapy
Drug: Flagyl — Metronidazole (Flagyl) 500 mg tid daily for 7 days in the non-bismuth quadruple therapy
  Other Names: Metronidazole
  Arms: Non-bismuth quadruple therapy

SUMMARY:
The Asian-Pacific Consensus Report has recommended that proton pump inhibitor (PPI)-clarithromycin-amoxicillin or metronidazole treatment for 7 to14 days is the first choice treatment for H pylori infection. As a general rule for the treatment of other infectious diseases, clinicians should prescribe therapeutic regimens that have a per-protocol eradication rate ≥ 90% for anti-H pylori therapy. However, the eradication rate of the standard triple therapy has generally declined to unacceptable levels (i.e., 80% or less) recently. The reasons for this fall in efficacy with time may relate to the increasing incidence of clarithromycin-resistant strains of H. pylori. Clarithromycin resistance is the major cause of eradication failure for stand triple therapy. Standard triple therapies should be abandoned in the areas with clarithromycin resistance ≥ 20% because the per-protocol eradication rates of standard therapies are often less than 85% and the intention-to-treat eradication rates are usually less than 80%..7-10 day non-bismuth containing quadruple therapy (Concomitant therapy) had been successful in the presence of clarithromycin resistance. Another novel treatment with 14-day high dose PPI and amoxicilin dual therapy could also attained >90 eradication rate in some studies. This novel treatment is simple and involved only two drugs and the most important of all is that amoxicillin resistance is still 0% in Taiwan . High dose PPI has been used in several studies for H. pylori eradication in order to increase the intra-gastric PH for optimal eradication So far, there is still unclear which one is the best first-line H. pylori eradication regimen with highest eradication rate and least adverse effects. We therefore design a randomized controlled trial to simultaneously assess the efficacy novel 14-day high dose dual therapy by comparing to the 7-day non-bismuth containing quadruple therapy in Taiwan and to investigate the host and bacterial factors predicting the treatment outcomes of eradication therapies.

DETAILED DESCRIPTION:
The Asian-Pacific Consensus Report has recommended that proton pump inhibitor (PPI)-clarithromycin-amoxicillin or metronidazole treatment for 7 to14 days is the first choice treatment for H pylori infection. As a general rule for the treatment of other infectious diseases, clinicians should prescribe therapeutic regimens that have a per-protocol eradication rate ≥ 90% for anti-H pylori therapy. However, the eradication rate of the standard triple therapy has generally declined to unacceptable levels (i.e., 80% or less) recently.[3-9] The reasons for this fall in efficacy with time may relate to the increasing incidence of clarithromycin-resistant strains of H. pylori. The main reasons for eradication failure for H pylori infection include antibiotic resistance, poor compliance and rapid metabolism of PPI. Clarithromycin resistance is the major cause of eradication failure for stand triple therapy. The rate of clarithromycin-resistant strains ranged from 49% (Spain) to 1% (Netherland) worldwide. Standard triple therapies should be abandoned in the areas with clarithromycin resistance ≥ 20% because the per-protocol eradication rates of standard therapies are often less than 85% and the intention-to-treat eradication rates are usually less than 80%. 7-10 day non-bismuth containing quadruple therapy (Concomitant therapy) had been successful in the presence of clarithromycin resistance. Another novel treatment with 14-day high dose PPI and amoxicilin dual therapy could also attained >90 eradication rate in some studies. This novel treatment is simple and involved only two drugs and the most important of all is that amoxicillin resistance is still 0% in Taiwan. High dose PPI has been used in several studies for H. pylori eradication in order to increase the intra-gastric PH for optimal eradication So far, there is still unclear which one is the best first-line H. pylori eradication regimen with highest eradication rate and least adverse effects. We therefore design a randomized controlled trial to simultaneously assess the efficacy novel 14-day high dose dual therapy by comparing to the 7-day non-bismuth containing quadruple therapy in Taiwan and to investigate the host and bacterial factors predicting the treatment outcomes of eradication therapies.

ELIGIBILITY:
Inclusion Criteria:

1. H. pylori-infected outpatients with endoscopically proven peptic ulcer diseases or gastritis.

Exclusion Criteria:

1. Previous H. pylori-eradication therapy
2. ingestion of antibiotics, bismuth, or PPIs within the prior 4 weeks
3. patients with allergic history to the medications used
4. patients with previous gastric surgery
5. the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
6. pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
The rates of H.pylori eradication | 6-8 weeks after treatment
  The primary outcome variables were the rates of eradication. Chi-square test with or without Yates correction for continuity and Fisher's exact test were used when appropriate to compare the major outcomes between groups. A P value less than 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Tai, MD, Principal Investigator — Kaohsiung Chang Gung Memorial Hospital,Taiwan
Locations (1):
- Wei-Chen Tai, Kaohsiung City, Taiwan